CLINICAL TRIAL: NCT05051540
Title: The Effect of Inelastic Compression System on Quality of Life in People With Chronic Venous Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hadar Lev-Tov, Assistant Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210807
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Chronic Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Inelastic Compression System Group (Experimental): Participants in this group will receive the inelastic compression wrap for daily use on their legs for 6 consecutive weeks.
  Interventions: Device: Sigvaris Compreflex Inelastic Compression Wrap

INTERVENTIONS:
Device: Sigvaris Compreflex Inelastic Compression Wrap — Compreflex compression system using wraps to apply compression of 30-40 mmHg.

SUMMARY:
The purpose of this protocol is to measure the effect of the use of an inelastic compression system (ICS) on quality of life (QOL) in patients with chronic venous insufficiency (CVI) who have demonstrated limited or no compliance with prescribed compression stockings or bandage wraps.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age 18 or older, able and willing to provide consent and agrees to comply with the study procedures
* Subject must have chronic venous insufficiency of stages C3, C4, or C5 according to the Clinical-Etiological-Anatomical-Pathophysiological (CEAP) classification system
* Not compliant with their currently prescribed compression system

Exclusion Criteria:

* Active malignancy other than non-melanoma skin cancer
* Study ulcer suspicious for cancer
* Subjects who are pregnant and/or breastfeeding
* In the opinion of the PI the subject cannot comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Lev-Tov, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inelastic Compression System Group
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Inelastic Compression System Group
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in the Quality of Life as Measured by CIVIQ-20
Description: Chronic Venous Disease Quality of Life Questionnaire (CIVIQ-20) consists of 20 multiple choice questions subdivided into four categories: psychology, pain, physical repercussions and social repercussions. The questionnaire has a total score ranging from 0 to 100 the lower score indicating greater quality of life.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inelastic Compression System Group
Number analyzed (Participants) | 30
score on a scale | 12.2 (21.06)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Inelastic Compression System Group
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT05051540/Prot_000.pdf